CLINICAL TRIAL: NCT04251104
Title: Effectiveness of the Level of Personal Relevance of Visual Autobiographical Stimuli in the Induction of Positive Emotions in Young and Older Adults: Study Protocol for a Randomized Controlled Trial
Brief Title: Effectiveness of Personal Relevance of Visual Autobiographical Stimuli in Positive Emotions Induction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government); European Regional Development Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SBPLY/19/180501/000181
Record Dates: First submitted 2020-01-16; First posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Emotion Regulation; Mood Induction; Autobiographical Memory; Ageing
Keywords: Images; personal relevance
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: This is an exploratory randomized controlled study to compare the effectiveness of three types of autobiographical stimuli, classified according to their level of personal relevance, in the induction of positive emotions resulting from the retrieval of specific positive autobiographical memories. The study sample will comprise a group of adults aged 65 years or over and a group of young adults aged between 18 and 35. Each participant will be assigned randomly to one of three parallel groups (high, medium and low personal relevance images). The allocation ratio will be 1:1:1.
Who Masked: Investigator
Masking Description: Psychologists responsible for participant recruitment will be blinded to the information about the group allocation. Due to the nature of the intervention neither participants nor psychologists responsible for the experimental phase can be blinded for the allocation, but the psychologist will be trained to decrease as much as possible her influence on the participants. For this, the psychologist will be provided with clear steps and norms to follow during the experimental intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Level of personal relevance of images (Experimental): This is an exploratory randomized controlled study to compare the effectiveness of three types of autobiographical stimuli, classified according to their level of personal relevance (high, medium and low), in the induction of positive emotions resulting from the retrieval of specific positive autobiographical memories. To this end, the investigators will use three types of images, classified according to their personal relevance: a) personal autobiographical photographs (high personal relevance); b) images of locations related to the participants' lives (medium personal relevance); and c) images from the Internation Affective Picture System (IAPS; low personal relevance).
  Interventions: Other: Images' personal relevance effectiveness in objective and subjective mood recovery
- Age (young and older adults comparison) (Other): To analyse any age-related differences in the effectiveness of the use of the three types of images to regulate emotion, the investigators will compare the efficacy of the three categories of pictures (high, medium and low relevance) in inducing positive mood states in a group of young adults (age range: 18-35 years) and a group of older adults (65 years or over).
  Interventions: Other: Images' personal relevance effectiveness in objective and subjective mood recovery

INTERVENTIONS:
Other: Images' personal relevance effectiveness in objective and subjective mood recovery — After completing the PANAS, the negative mood induction phase (viewing a film clip) phase will begin. Before this phase, the participants will be encouraged to experience the feelings generated by the clip as intensely as possible. After viewing the film clip, participants will be asked to complete the PANAS again in order to assess the effectiveness of the negative mood induction procedure.
  Following the negative mood induction phase, the emotional recovery phase will be initiated, in which the participants will look at a total of six pictures previously selected according to their experimental condition in order to generate specific positive autobiographical memories. At the end of this phase, participants will once more complete the PANAS in order to assess the effectiveness of the emotional recovery.

SUMMARY:
Background: The ability to retrieve specific memories is a cognitive and emotional protective factor. Among the most effective techniques to generate autobiographical memories is the use of audio-visual stimuli, particularly images. Developing and improving techniques that facilitate the generation of such memories could be highly effective in the prevention of depressive symptoms, especially in the elderly population. The aim of the present study is to examine how the level of personal relevance of pictures as autobiographical memory cues to induce positive emotions may affect an individual's emotion regulation.

Methods: The participants, 120 older adults aged 65 and over and 120 young adults aged between 18 and 35, of both sexes and without depressive symptoms, will be induced to a negative mood state by means of viewing a film clip. Following the negative mood induction, the participants will be shown positive images according to experimental group to which they were randomly assigned (high personal relevance: personal autobiographical photographs; medium personal relevance: pictures of favourite locations associated with specific positive autobiographical memories; and low personal relevance: positive images from the International Affective Picture System). The investigators will analyse the differences in subjective (responses to questionnaires) and objectives measures (EEG signal, heart rate variability and electrodermal activity) between the groups before and after the induction of negative affect and following the recall of positive memories.

Discussion: The use of images associated with specific positive autobiographical memories may be an effective input for inducing positive mood states, which has potentially important implications for their use as a cognitive behavioural technique to treat emotional disorders, such as depression, which are highly prevalent among older adults.

ELIGIBILITY:
Inclusion Criteria:

1. Older adults will present no symptoms of cognitive impairment. The self-administered Test Your Memory (TYM) will be used to assess cognitive performance [79,80].
2. Absence of depressive symptomatology, which will be assessed using the Patient-Reported Outcomes Measurement Information System-Depression [81].
3. Given the high comorbidity between anxiety and depression [82,83], it was decided that both young and older participants should present no symptoms of anxiety. This will be assessed using the Patient-Reported Outcomes Measurement Information System-Anxiety [81].
4. No sensory deficits that might impact performance in the experiment and the psychological tests.
5. Sufficient literacy skills to understand the instructions for the experiment and the psychological tests.
6. Signed informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study will include both men and women, aiming for a proportion of at least 40% and 60%.
Enrollment: 240 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Mood state measures: Positive and Negative Affect Schedule (PANAS) | Positive and Negative Affect scales are administered before and after the negative mood induction and before the emotional recovery. The experimental task lasts 25 min. Each scale scores from 10 to 50. Higher scores mean higher affect.
  Assessment of positive and negative affect during the experimental phase
Hemispheric frontal asymmetry in EEG activity | Fast Fourier transformation will be applied to an EEG epoch consisting of the time windows of 30 s each after the onset of the stimulus (film and images) during the experimental task (maximum duration 25 minutes)
  Left frontal (F3, F7, FC5) and right frontal (F4, F8, FC6) electrode pools will be formed by averaging the frequency distributions of these signals
EEG power in delta band | Fast Fourier transformation will be applied to an EEG epoch consisting of the time windows of 30 s each after the onset of the stimulus (film and images) during the experimental task (maximum duration 25 minutes)
  The mean magnitud of delta frequency band activity will be calculated for each participant during each event type (film and images).
EEG power in theta band | Fast Fourier transformation will be applied to an EEG epoch consisting of the time windows of 30 s each after the onset of the stimulus (film and images) during the experimental task (maximum duration 25 minutes)
  The mean magnitud of theta frequency band activity will be calculated for each participant during each event type (film and images).
EEG power in alpha band | Fast Fourier transformation will be applied to an EEG epoch consisting of the time windows of 30 s each after the onset of the stimulus (film and images) during the experimental task (maximum duration 25 minutes)
  The mean magnitud of alpha frequency band activity will be calculated for each participant during each event type (film and images).
EEG power in beta band | Fast Fourier transformation will be applied to an EEG epoch consisting of the time windows of 30 s each after the onset of the stimulus (film and images) during the experimental task (maximum duration 25 minutes)
  The mean magnitud of beta frequency band activity will be calculated for each participant during each event type (film and images).
EEG power in gamma band | Fast Fourier transformation will be applied to an EEG epoch consisting of the time windows of 30 s each after the onset of the stimulus (film and images) during the experimental task (maximum duration 25 minutes)
  The mean magnitud of gamma frequency band activity will be calculated for each participant during each event type (film and images).
Electrodermal activity (EDA) or skin conductance (SC) | Skin conductance is registered during all the experimental task (maximum duration: 25 minutes).
  SC morphology is the result of two independent components: a fast-changing skin conductance response (SCR), overlapped with a slowly changing skin conductance level component (SCL). The SCL component ranges from 0Hz to 0.05Hz, while SCR ranges from 0.05Hz to 1.5 Hz. Each SC signal will be filtered by applying a 1.5Hz cut-off low-pass FIR filter to decrease noise generated during the acquisition. The data series will first be divided into equal segments lasting five seconds and the mean of each segment will be recorded for subsequent analysis.
Heart rate variability (HRV) | HRV is registered during all the experimental task (maximum duration: 25 minutes)..
  Cardiovascular variables will be measured through blood volume pressure (BVP). Alternations of the BVP waveform are highly correlated with heart ventricular depolarization and repolarization, thus being suitable to measure heart rhythm. Once data are acquired, BVP signals will be processed to reduce noise. After that, interbeat intervals (IBIs) will be derived from the peak-data series. The IBI data series will be transformed to obtain the heart rate (HR) measured in beats per minute (BPM). Then, the HR metric will be partitioned into five-second equally-separated segments.

REFERENCES:
- [Derived] Fernandez D, Ros L, Sanchez-Reolid R, Ricarte JJ, Latorre JM. Effectiveness of the level of personal relevance of visual autobiographical stimuli in the induction of positive emotions in young and older adults: pilot study protocol for a randomized controlled trial. Trials. 2020 Jul 20;21(1):663. doi: 10.1186/s13063-020-04596-5. PMID 32690050